CLINICAL TRIAL: NCT01803334
Title: Impact of Marking Surgical Incision Size and Location on the Patient's Abdomen During Preoperative Counseling in Minimally Invasive Gynecologic Surgery. A Randomized Control Trial.
Brief Title: Impact of Marking Surgical Incision on Patient's Abdomen
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants could be enrolled and so the PI decided to close the study. No participants completed the study
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 322259
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Surgical Procedure
Keywords: surgical incision; laparoscopy; pain
MeSH Terms: conditions — Surgical Wound; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marking abdomen (Experimental): If the patient is randomized to the marking the abdomen group (study group) she will then have the anticipated incision needed to place the trocars during her surgery marked on her abdomen by the surgeon attending physician involved in the patient care during the preoperative counseling visit.
  Interventions: Other: Marking abdomen
- Control (No Intervention): If she is randomized to the control group, then she will undergo traditional preoperative counseling by the same team without marking the abdomen.

INTERVENTIONS:
Other: Marking abdomen — If the patient is randomized to the marking the abdomen group (study group) she will then have the anticipated incision needed to place the trocars during her surgery marked on her abdomen by the surgeon attending physician involved in the patient care during the preoperative counseling visit.
  Arms: Marking abdomen

SUMMARY:
This is a study looking at patient's satisfaction with incision site and location after undergoing minimally invasive gynecologic surgery. (Laparoscopy) The study group will have the anticipated incision marked with a washable marker on their abdomen. The control group will have preoperative counselling as usual. After surgery, will assess patient's satisfaction with the incision scar.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled trial examining the impact of marking the patient abdomen at the time of the preoperative visit on patient's satisfaction with scar appearance and symptoms, and pain at the incision site after undergoing minimally invasive gynecologic surgery for benign conditions.

We hypothesize that preoperative marking and instruction about incision expectations will improve patient's postoperative satisfaction with scar appearance and symptoms as well as decrease incision site pain compared to traditional preoperative counseling.

Patients that will undergo laparoscopic surgical intervention will be identified. The patient will be randomized into two groups: preoperative marking the abdomen versus conventional preoperative counseling.

If the patient is randomized to the marking the abdomen group (study group) she will then have the anticipated incision needed to place the trocars during her surgery marked on her abdomen by the surgeon attending physician involved in the patient care during the preoperative counseling visit. If she is randomized to the control group, then she will undergo traditional preoperative counseling by the same team without marking the abdomen.

After completed the surgery, information regarding type of surgery, reason for the procedure, estimated blood loss, surgical length, complications, location and size of abdominal incisions made on the patient's abdomen will be collected. Then at the 6 weeks post op visit, patient's satisfaction with the incision scar will be evaluated with a validated patient scar assessment questionnaire form and by one 5 point Likert scale question used in previous studies. The pain at rest at the incision site will be evaluated by a Visual Analog Pain Scale (VAS). Patients will also be asked to evaluate their generalized pain using a modified McGill Present Pain Intensity Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 89
2. Diagnosed with a benign surgical pathology
3. Patient scheduled for elective minimally invasive gynecologic surgery

Exclusion Criteria:

1. Have a diagnosis of gynecologic cancer
2. History of prior laparoscopic surgery
3. Emergency surgery
4. Inability to provide informed consent
5. Unable to follow up in the office for post operative visits
6. Skin hypersensitivity or allergy to marker dye
7. Positive pregnancy test

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07-08 (Actual); Study Completion 2013-07-08 (Actual)

PRIMARY OUTCOMES:
Patient's expectation and satisfaction with incision scar will be evaluated with the patient scar assessment questionnaire and a 5 points Likert type scale question. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose A carugno, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Orlando, Florida, United States